CLINICAL TRIAL: NCT06740799
Title: A Phase 1, Multicenter, Open-Label, Single-Dose Study to Assess the Pharmacokinetics, Safety and Tolerability of Quizartinib in Subjects With Severe Impaired Hepatic Function
Brief Title: Assessment of Quizartinib Pharmacokinetic in Subjects With Severe Hepatic Impairment
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Daiichi Sankyo (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AC220-163
Record Dates: First submitted 2024-12-13; First posted 2024-12-18 (Actual); Last update posted 2025-10-14 (Actual); Status verified 2025-10

CONDITIONS: Hepatic Impairment
Keywords: quizartinib
MeSH Terms: interventions — quizartinib

STUDY DESIGN:
Masking Description: No masking,
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Severe HI (Experimental): Participants will receive a single oral dose of 30 mg quizartinib
  Interventions: Drug: Quizartinib
- Control Group (Experimental): Healthy participants will receive a single oral dose of 30 mg quizartinib
  Interventions: Drug: Quizartinib

INTERVENTIONS:
Drug: Quizartinib — Participants will receive a single oral dose of 30 mg
  Other Names: Test Product; VANFLYTA®

SUMMARY:
This study will evaluate and compare the PK in subjects with severe HI to that of matched healthy control subjects with normal hepatic function.

DETAILED DESCRIPTION:
This is a clinical pharmacology study with 2 cohorts (subjects with severe HI by Child-Pugh criteria and matched healthy control subjects) to evaluate the PK, safety, and tolerability of a single oral dose of 30 mg quizartinib in otherwise healthy subjects with severe HI (as defined by Child-Pugh criteria). This study is planned to be conducted at up to 3 sites in the US, which use Child-Pugh criteria.

ELIGIBILITY:
Key Inclusion Criteria:

1. Voluntarily consents to participate in this study and provides written informed consent before the start of any study-specific procedures.
2. Male and female subjects 18 to 75 years of age (inclusive), with a body mass index (BMI) of 18 kg/m2 to 37 kg/m2 (inclusive) with a minimum body weight of 40 kg at Screening.
3. In females, documented surgical sterilization (ie, documented hysterectomy, bilateral tubal ligation, or bilateral salpingo-oophorectomy, Essure® with hysterosalpingogram [documentation to confirm tubal occlusion 12 weeks after procedure]), postmenopausal status for at least 1 year (follicle stimulating hormone [FSH] > 40 mIU/mL serum and estradiol <40 pg/mL [<147 pmol/L] at Screening), or agreement to have a sterile male partner, or agreement to use 1 of the means of contraception from Screening until 7 months after the dose of quizartinib 4. In females, agreement to not retrieve eggs/ova via assisted reproductive technology (ART) either for their own use or donation while on the study or for 7 months after the last dose of study drug, whichever is later.

5. In males, documented surgical sterilization, sexual abstinence, or agreement to use 1 of the means of contraception from Screening until 4 months after the dose of quizartinib 6. In males, agreement to avoid sperm donation for 4 months after the dose of quizartinib

Key Exclusion:

1. Any serious and/or unstable pre-existing medical, psychiatric disorder, or other conditions (including lab abnormality except hepatic impairment) that could interfere with safety, obtaining informed consent, compliance to the study procedures, or the validity of the study results.
2. In the opinion of the investigator, history of a clinically significant illness within 4 weeks prior to administration of quizartinib.
3. Subjects with primary biliary cirrhosis or primary sclerosing cholangitis.
4. Subjects with history of Gilbert's syndrome.
5. Presence or history of clinically severe adverse reaction to any drug or known hypersensitivity to any of the ingredients (including inactive ingredients) of quizartinib.
6. History of stomach or intestinal surgery or resection that would potentially alter absorption and/or excretion of orally administered drugs (with the exception of appendectomy, hernia repair, and/or cholecystectomy).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2024-09-30 (Actual); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
Pharmacokinetic Parameter: Cmax | From day of first dose, Day 1, through Day 29
  Maximum concentration, determined directly from individual concentration-time data
Pharmacokinetic Parameter: Tmax | From day of first dose, Day 1, through Day 29
  Time of the maximum concentration
Pharmacokinetic Parameter: AUClast | From day of first dose, Day 1, through Day 29
  Area under the concentration-time curve from time-zero to the time of the last quantifiable concentration; calculated using the linear up log down
Pharmacokinetic Parameter: AUCinf | From day of first dose, Day 1, through Day 29
  Area under the concentration-time curve from time-zero extrapolated to infinity
Pharmacokinetic Parameter: t1/2 | From day of first dose, Day 1, through Day 29
  The observed terminal half-life

SECONDARY OUTCOMES:
Treatment Emergent Adverse Events | From day of first dose, Day 1, up to 30 days after Day 29
  TEAEs are defined as new AEs that occur after the first dose of study drug

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Leader, Study Director — Daiichi Sankyo
Locations (3):
- United States (3):
  - Clinical Pharmacology of Miami, LLC, Miami, Florida
  - Advanced Pharma, Miami, Florida
  - GCP Research, St. Petersburg, Florida

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) on completed studies and applicable supporting clinical trial documents may be available upon request at https://vivli.org/. In cases where clinical trial data and supporting documents are provided pursuant to our company policies and procedures, Daiichi Sankyo will continue to protect the privacy of our clinical trial participants. Details on data sharing criteria and the procedure for requesting access can be found at this web address: https://vivli.org/ourmember/daiichi-sankyo
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Completed studies that has reached a global end or completion with all data set collected and analyzed, and for which the medicine and indication have received European Union (EU) and United States (US), and/or Japan (JP) marketing approval on or after 01 January 2014 or by the US or EU or JP Health Authorities when regulatory submissions in all regions are not planned and after the primary study results have been accepted for publication.
Access Criteria: Formal request from qualified scientific and medical researchers on IPD and clinical study documents on completed clinical trials supporting products submitted and licensed in the United States, the European Union and/or Japan from 01 January 2014 and beyond for the purpose of conducting legitimate research. This must be consistent with the principle of safeguarding study participants' privacy and consistent with provision of informed consent.
URL: https://vivli.org/ourmember/daiichi-sankyo/